CLINICAL TRIAL: NCT00756925
Title: Exploring Gender Differences in the Neural Substrates of Stress Induced Drug Craving
Brief Title: Gender and Neural Substrates of Stress and Craving
Status: Completed | Type: Observational
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Megan Moran-Santa Maria, Assistant Professor, Medical University of South Carolina
Other Study IDs: HR18441
Record Dates: First submitted 2008-09-18; First posted 2008-09-22 (Estimated); Last update posted 2018-05-07 (Actual); Status verified 2018-05

CONDITIONS: Cocaine Dependence
Keywords: CRH; cocaine; functional magnetic resonance imaging; gender differences
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — corticorelin ovine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Cocaine dependent females
  Interventions: Drug: Acthrel
- 2: Cocaine dependent males
  Interventions: Drug: Acthrel

INTERVENTIONS:
Drug: Acthrel — 1 ug/kg, i.v., 1 minute

SUMMARY:
Cocaine dependence is an insidious disease underscored by a powerful proclivity to relapse despite an individual's ability to recognize the deleterious consequences of continued drug use. To date, there are only a limited number of treatments, and no FDA approved medications for the treatment of cocaine dependence. Attempts to find reliable and successful treatments for cocaine dependence may be marred by gender differences in brain chemistry, structure, and function that are manifested as drug craving and relapse. For example, cues, drug exposure, and stress promote relapse, yet females appear be more susceptible to stress induced relapse, while males may be more susceptible to cue induced relapse. Therefore identifying the neural substrates involved in processing the valence of internal and external stimuli may provide further insight into cocaine dependence and provide more effective therapeutic strategies aimed at preventing relapse.

Corticotropin releasing hormone (CRH) is a pharmacological activator of the hypothalamic pituitary adrenal (HPA) axis, and has been implicated in stress induced drug relapse. Corticotropin releasing hormone receptors are located at extrahypothalamic brain nuclei that have been implicated in determining the significance of both internal (somatic) and external (environmental) stimuli. The primary directive of this pilot project is to utilize functional magnetic resonance imaging (fMRI) to identify possible brain nuclei associated with with stress induced drug craving in cocaine dependent females.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65
2. Right-handed
3. Males and females meeting criteria for cocaine dependence (DSM-IV), within the past three months (current).
4. Subjects must be able to provide informed consent and function at an intellectual level sufficient to allow accurate completion of all assessment instruments.
5. Subjects must consent to remain abstinent from all drugs of abuse (except nicotine) for a three-day period immediately prior to the GCRC admission. Nicotine dependence can affect HPA function therefore it would be ideal to exclude subjects with nicotine use. Because of the comorbidity of cocaine and nicotine dependence, this would seriously compromise the feasibility of recruitment. Alcohol has also been known to affect HPA function, however to enhance recruitment efforts, individuals with alcohol dependence or abuse will be included in the study if they do not require medically supervised detoxification.
6. Participants must have a negative breathalyzer, urine drug screen.
7. Subjects must consent to outpatient admission to the GCRC

Exclusion Criteria:

1. Subjects with evidence of or a history of significant hematological, endocrine, cardiovascular, pulmonary, renal, gastrointestinal, or neurological disease including diabetes, as these conditions may affect HPA axis function.
2. Subjects with any liver function test of greater than two times normal, as compromised liver function can interfere with HPA axis activity.
3. Subjects with Addison's disease, Cushing's disease or other diseases of the adrenal cortex likely to affect HPA axis function.
4. Subjects with a history of or current psychotic disorder or bipolar affective disorder as these may interfere with HPA function.
5. Subjects with current major depressive disorder or post-traumatic stress disorder as these disorders are associated with characteristic changes in HPA axis function.
6. Subjects receiving synthetic glucocorticoid therapy, any exogenous steroid therapy, or treatment with other agents, that interfere with HPA axis function within one month of the time of testing.
7. Subjects taking opiates, opiate antagonists, or benzodiazepines. (Subjects who have been maintained on SSRI's, anticonvulsants, or antipsychotics (for sleep only) for more than 8 weeks or longer are NOT excluded).
8. Subjects with any acute illness or fever as this may affect HPA axis activity. Individuals who otherwise meet study criteria will be rescheduled for evaluation for participation.
9. Subjects who are > 30% over ideal weight or have a BMI greater than 30 will be considered for study participation based on the clinical judgment of study staff.
10. Subjects who are unwilling to maintain abstinence from alcohol and other drugs of abuse (except nicotine) for two days prior to the stress task procedure.
11. Persons with ferrous metal implants or pacemaker since fMRI will be used.
12. Subjects that are claustrophobic

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 20 cocaine dependent subjects (10 cocaine dependent females and 10 cocaine dependent males) will be enrolled in the study. Inclusion/exclusion criteria are listed in Section E, Human Subjects. Cocaine subjects will be matched for age and nicotine dependence. Women taking birth control pills, or Depo Provera (medroxyprogesterone acetate) will be excluded from study participation.
  Subjects will be recruited through the use of flyers, advertisements on the MUSC website, MUSC broadcast messages, advertisement in local newspapers and weeklies, and similar ongoing studies within the Clinical Neuroscience Division.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2009-02; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Neurosciences Division-Medical University of South Carolina, Charleston, South Carolina, United States